CLINICAL TRIAL: NCT06115460
Title: The Impact of Sitagliptin as an Add on Therapy With Closed Loop Control in Adolescents With Type 1 Diabetes Mellitus and Diabetic Nephropathy
Brief Title: The Impact of Sitagliptin as an Add on Therapy With Closed Loop Control in Adolescents With Diabetic Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Nancy Samir Elbarbary, Prof. of Pediatrics, Ain Shams University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ain Shams University202388
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Type 1 Diabetic Nephropathy
Keywords: Type 1 diabetes; Diabetic nephropathy; Sitagliptin; Time in Range; Advanced hybrid closed system; Stromal cell-derived factor-1 (SDF-1)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral sitagliptin 50 mg supplementation for three months (Active Comparator): Intervention group includes: adolescents with diabetic nephropathy on advanced hybrid closed loop system receiving oral sitagliptin 50 mg for three months on a daily basis
  Interventions: Drug: oral sitagliptin supplementation
- Control group ( No intake of oral sitagliptin 50 mg supplementation for three months) (No Intervention): Control group includes: adolescents with diabetic nephropathy on advanced hybrid closed loop system who did not take oral sitagliptin 50 mg for three months on a daily basis

INTERVENTIONS:
Drug: oral sitagliptin supplementation — oral sitagliptin supplementation for three months
  Arms: Oral sitagliptin 50 mg supplementation for three months

SUMMARY:
Diabetic nephropathy (DN) is one of the most frequent microvascular complications of diabetes mellitus, affecting 25 to 40% of patients with type 1 diabetes (T1DM). Early diagnosis, appropriate patient follow-up and treatment are essential to improve the outcomes. There is a need for improvements in insulin therapy for people with T1DM as the majority of patients are struggling to achieve glycemic targets. Technological advancements and oral adjuncts to insulin therapies are starting to be licensed for the use of people with T1DM.

Dipeptidyl peptidase-4 (DPP-4), a multifunctional serine protease with a dual function (regulatory protease and binding protein), can modulate inflammation and immune cell-mediated β-cell destruction. DPP-4 degrades the peptide hormones glucagon-like peptide 1 (GLP-1) and gastric inhibitory peptide (GIP). Several studies have suggested that the upregulated DPP-4 activity is correlated with T1DM pathophysiology.

DETAILED DESCRIPTION:
Evidence from preclinical investigation suggests that DPP-4 inhibition may have beneficial effects on various metabolic indicators in diabetes. DPP-4 inhibitors, such as sitagliptin, have been widely used as outstanding blood glucose-dependent antidiabetic agents for patients with type 2 diabetes(T2DM). DPP-4 inhibitors have a lowering effect on the glycemic level and were not associated with increasing incidence of adverse events. The reno-protective effects of DPP-4 inhibition in diabetic nephropathy could be a consequence of the antidiabetic actions of DPP-4 inhibitors.

A second-generation advanced hybrid closed loop ( AHCL) system has been developed to further improve glycemic control and usability, with adjustable target glucose and automated correction boluses. This system provides proportional integral derivate (PID) algorithm with insulin feedback with adaptive insulin limits and model based auto-corrections located on the pump. Sitagliptin demonstrated an overall decrease in blood glucose concentrations in adults with T1DM when used as an adjunct therapy with an insulin only closed loop (CL) system.

Stromal cell-derived factor-1 (SDF-1) is ubiquitously expressed in diverse organs and has multiple functions. SDF-1 is cleaved and inactivated by the DPP-4 enzyme. The DPP-4 enzyme is highly expressed in the kidney. It has been suggested that renal SDF-1 upregulation by DPP-4 inhibition produces multiple protective actions on the diabetic kidney.

In view of these data, the investigators assessed the impact of sitagliptin as add on therapy with closed loop control in adolescents with T1DM on glycemic control, diabetic nephropathy and SDF-1 as a marker for nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* T1DM patients aged 12-18 years with at least 5 years disease duration defined according to the criteria of International Society for Pediatric and Adolescent Diabetes (ISPAD) .
* Patients on insulin pump therapy using Medtronic advanced hybrid closed system (Medtronic, Northridge, USA) with Guardian™ 3 sensor or Guardian™ 4 sensor and Guardian link transmitter initiated at least 6 months before the study, patients with minimum daily insulin requirement of more than 8 units, willingness and ability to adhere to the study protocol, and access to the internet as well as a computer system that met requirements for uploading the study pump data.
* Active diabetic nephropathy in the form of microalbuminuria (urinary albumin excretion ) 30-299 mg/g creatinine in two of three samples over a 3- to 6-months period despite angiotensin converting enzyme inhibitors).
* Hemoglobin A1c (HbA1c) ≤8.5%.
* Patients on regular visits to clinic.

Exclusion Criteria:

* patients with other diabetic microvascular complications (neuropathy or retinopathy) or with macrovascular complications.
* Patients with history of liver disease or any disorder likely to impair liver functions or elevated liver enzymes.
* Patients with any evidence of renal impairment due to causes other than diabetes.
* Patients with hypertension.
* Hepatitis virus infection (B or C) or any evidence of infection
* Participation in a previous investigational drug study within 3 months preceding screening.
* Hypoglycemic unawareness or recurrent severe hypoglycemic episodes in the last 6 months prior to recruitment.
* Recurrent diabetic ketoacidosis (DKA) (more than 2 episodes in the previous 6 months).
* Taking other oral hypoglycemic medications which could affect blood glucose.
* Patients with known allergy to sitagliptin.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Time in range | 3 months
  Change in Time in range (TIR) in intervention group in comparison to control group

SECONDARY OUTCOMES:
Level of microalbuminuria | 3 months
  Change in microalbuminuria level in intervention group in comparison to control group
Level of Stromal cell-derived factor-1 (SDF-1) | 3 months
  Change in Stromal cell-derived factor-1 (SDF-1)in intervention group in comparison to control group

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy Elbarbary, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
All data are available upon request

REFERENCES:
- [Background] Zhong J, Rajagopalan S. Dipeptidyl Peptidase-4 Regulation of SDF-1/CXCR4 Axis: Implications for Cardiovascular Disease. Front Immunol. 2015 Sep 25;6:477. doi: 10.3389/fimmu.2015.00477. eCollection 2015. PMID 26441982
- [Background] Weisman A, Bai JW, Cardinez M, Kramer CK, Perkins BA. Effect of artificial pancreas systems on glycaemic control in patients with type 1 diabetes: a systematic review and meta-analysis of outpatient randomised controlled trials. Lancet Diabetes Endocrinol. 2017 Jul;5(7):501-512. doi: 10.1016/S2213-8587(17)30167-5. Epub 2017 May 19. PMID 28533136
- [Background] Williams-Herman D, Engel SS, Round E, Johnson J, Golm GT, Guo H, Musser BJ, Davies MJ, Kaufman KD, Goldstein BJ. Safety and tolerability of sitagliptin in clinical studies: a pooled analysis of data from 10,246 patients with type 2 diabetes. BMC Endocr Disord. 2010 Apr 22;10:7. doi: 10.1186/1472-6823-10-7. PMID 20412573
- [Background] Garg SK, Weinzimer SA, Tamborlane WV, Buckingham BA, Bode BW, Bailey TS, Brazg RL, Ilany J, Slover RH, Anderson SM, Bergenstal RM, Grosman B, Roy A, Cordero TL, Shin J, Lee SW, Kaufman FR. Glucose Outcomes with the In-Home Use of a Hybrid Closed-Loop Insulin Delivery System in Adolescents and Adults with Type 1 Diabetes. Diabetes Technol Ther. 2017 Mar;19(3):155-163. doi: 10.1089/dia.2016.0421. Epub 2017 Jan 30. PMID 28134564
- [Background] Bergenstal RM, Nimri R, Beck RW, Criego A, Laffel L, Schatz D, Battelino T, Danne T, Weinzimer SA, Sibayan J, Johnson ML, Bailey RJ, Calhoun P, Carlson A, Isganaitis E, Bello R, Albanese-O'Neill A, Dovc K, Biester T, Weyman K, Hood K, Phillip M; FLAIR Study Group. A comparison of two hybrid closed-loop systems in adolescents and young adults with type 1 diabetes (FLAIR): a multicentre, randomised, crossover trial. Lancet. 2021 Jan 16;397(10270):208-219. doi: 10.1016/S0140-6736(20)32514-9. PMID 33453783
- [Background] Ho TK, Shiwen X, Abraham D, Tsui J, Baker D. Stromal-Cell-Derived Factor-1 (SDF-1)/CXCL12 as Potential Target of Therapeutic Angiogenesis in Critical Leg Ischaemia. Cardiol Res Pract. 2012;2012:143209. doi: 10.1155/2012/143209. Epub 2012 Feb 22. PMID 22462026
- [Derived] Elbarbary NS, Ismail EA, El-Hamamsy MH, Ibrahim MZ, Elkholy AA. The DPP-4 inhibitor sitagliptin improves glycaemic control and early-stage diabetic nephropathy in adolescents with type 1 diabetes using the MiniMed 780G advanced hybrid closed-loop system: a randomised controlled trial. Diabetologia. 2024 Dec;67(12):2637-2649. doi: 10.1007/s00125-024-06265-7. Epub 2024 Sep 14. PMID 39271520